CLINICAL TRIAL: NCT01673386
Title: A Phase 2 Randomized, Double-Blind, Crossover, Controlled, Multi-Center Subject Preference Study of Tivozanib Hydrochloride Versus Sunitinib in the Treatment of Subjects With Metastatic Renal Cell Carcinoma
Brief Title: A Subject Treatment Preference Study of Tivozanib Versus Sunitinib in Subjects With Metastatic RCC
Acronym: TAURUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor
Sponsor: AVEO Pharmaceuticals, Inc. (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AV-951-12-205
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Tivozanib hydrochloride; renal cell carcinoma; subject preference; quality of life
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — tivozanib; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tivozanib Hydrochloride (Experimental): 1.5 mg oral tivozanib hydrochloride daily on a 3 weeks on/1 week off schedule for 12 weeks, followed by 50 mg oral sunitinib daily on a 4 weeks on/2 weeks off schedule for 12 weeks.
  Interventions: Drug: Tivozanib
- Sunitinib (Active Comparator): 50 mg oral sunitinib daily on a 4 weeks on/2 weeks off schedule for 12 weeks, followed by 1.5 mg oral tivozanib hydrochloride daily on a 3 weeks on/1 week off schedule for 12 weeks.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Tivozanib
  Other Names: Tivozanib Hydrochloride
  Arms: Tivozanib Hydrochloride
Drug: Sunitinib
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
Randomized, double-blind, 2-arm crossover study comparing tivozanib hydrochloride and sunitinib in subjects with metastatic RCC who have received no prior systemic therapy for Renal Cell Carcinoma (RCC).

DETAILED DESCRIPTION:
This is a randomized, double-blind, 2-arm crossover study comparing tivozanib hydrochloride and sunitinib in subjects with metastatic RCC who have received no prior systemic therapy for Renal Cell Carcinoma (RCC). Approximately 160 subjects will be stratified for ECOG score (0 vs 1) and histology (clear cell vs non-clear cell) and then will be randomized 1:1 to 1 of 2 treatment arms. The study consists of two 12-week treatment periods with a 1-week washout in between. Subjects will receive double-blind (over-encapsulated) tivozanib hydrochloride and sunitinib sequentially. The study is designed to compare subject treatment preference, as well as overall safety and tolerability, frequency of dose modifications and kidney-specific health outcomes/QoL.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable mRCC
* Histologically or cytologically confirmed RCC of any histology
* Subjects with or without prior nephrectomy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Any prior systemic therapy for treatment of mRCC (including investigational or licensed drugs that target VEGF or VEGF receptors/pathway, or are mammalian target of rapamycin [mTOR] inhibitors)
* Central nervous system malignancies or metastases
* Significant hematologic, gastrointestinal, thromboembolic, vascular, bleeding, or coagulation disorders
* Significant serum chemistry or urinalysis abnormalities
* Significant cardiovascular disease, including symptomatic left ventricular ejection fraction or baseline LVEF of ≤ institutional lower limit of normal, uncontrolled hypertension, myocardial infarction or severe angina within 6 months prior to administration of first dose of study drug, history of class III or IV congestive heart failure, or history of serious ventricular arrhythmia, cardiac arrhythmias, or coronary or peripheral bypass graft within 6 months of screening
* Corrected QT interval (QTc) of >480 msec using Bazett's formula
* Currently active second primary malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Needle, MD, Study Chair — AVEO Pharmaceuticals, Inc.
Locations (38):
- United States (15):
  - Los Angeles, California
  - Albany, Georgia
  - Atlanta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Worcester, Massachusetts
  - Minneapolis, Minnesota
  - New York, New York
  - Columbus, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - San Antonio, Texas
  - Madison, Wisconsin
- Belgium (2):
  - Antwerp
  - Brussels
- France (4):
  - Bordeaux
  - Caen
  - Lyon
  - Paris
- Germany (5):
  - Berlin
  - Hamburg
  - Hanover
  - Heidelberg
  - Munich
- Italy (3):
  - Aviano
  - Pavia
  - Rome
- Spain (4):
  - Barcelona
  - Madrid
  - Pamplona
  - Valencia
- United Kingdom (5):
  - Glasgow, Scotland
  - Swansea, Wales
  - Cambridge
  - London
  - Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aveo Pharmaceuticals, Inc. official web page — http://www.aveooncology.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All screening assessments were performed within 28 days prior to the first dose of study drug. All subjects were recruited as per the inclusion and exclusion criteria.
Groups:
- Tivozanib First, Then Sunitinib: Subject randomized to this arm received 1.5 mg oral tivozanib hydrochloride (drug 1) daily on a 3 weeks on/1 week off schedule for 12 weeks, followed by 50 mg oral sunitinib (drug 2) daily on a 4 weeks on/2 weeks off schedule for 12 weeks.
- Sunitinib First, Then Tivosanib: Subject randomized to this arm received 50 mg oral sunitinib (drug 1) daily on a 4 weeks on/2 weeks off schedule for 12 weeks, followed by 1.5 mg oral tivozanib hydrochloride (drug 2) daily on a 3 weeks on/1 week off schedule for 12 weeks.
Period: Overall Study
Arm/Group | Tivozanib First, Then Sunitinib | Sunitinib First, Then Tivosanib
Started | 27 | 31
Completed | 2 (Of 2 subjects, 1 subject discontinued tivozanib early, completed planned treatment with sunitinib.) | 4 (Of 4 subjects, 3 subjects discontinued sunitinib early, completed planned treatment with tivozanib.)
Not Completed | 25 | 27
Not completed — Study terminated by sponsor | 16 | 22
Not completed — Adverse Event | 5 | 2
Not completed — Progressive disease | 4 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects randomized to Arm 1, received 1.5 mg oral tivozanib daily on a 3 week on/1 week off schedule for 12 weeks (3 cycles) followed by 50 mg oral sunitinib daily on a 4 week on/2 week off schedule for 12 weeks (2 cycles). Subjects randomized to Arm 2, received 50 mg oral sunitinib daily on a 4 week on/2 weeks off schedule for 12 weeks followed by 1.5 mg oral tivozanib daily on a 3 week on/1 week off schedule.
Arm/Group | Overall Study
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 32
Age, Continuous [Median (Full Range); unit: years] | 65.5 [38 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 56
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Prefer Tivozanib Hydrochloride or Sunitinib
Description: The study was terminated prior to completing enrollment; due to low enrollment, no data was collected for this outcome measure.
Time Frame: Up to 25 weeks
Population: The study was terminated prior to completing enrollment; due to low enrollment, no data was collected for this outcome measure.
Groups:
- Tivozanib: Tivozanib hydrochloride 1.5 mg was administered orally to the randomized subjects first in arm 1 and second in arm 2.
- Sunitinib: Sunitinib 50 mg was administered orally to the randomized subjects first in arm 2 and second in arm 1.
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Subjects With AEs and SAEs
Description: Number of subjects with serious and non-serious adverse events.
Time Frame: Up to 25 weeks
Population: Descriptive statistical analyses were performed for a limited set of data (disposition, demographics, and adverse events).
Measure: Count of Participants; unit: Participants
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 38 | 41
Participants
  At least one AE | 35 | 40
  At least one treatment-related AE | 33 | 38
  At least one serious AE (SAE) | 6 | 7
  At least one treatment-related SAE | 1 | 3
  At least one AE leading to drug withdrawal | 3 | 8
  At least one AE with outcome of death | 2 | 1

3. Secondary Outcome: Number of Subjects With Dose Reductions
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Subjects With Dose Interruptions
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Subjects With Grade 3/4 Hematology Abnormalities
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Subjects With Grade 3/4 Chemistry Abnormalities
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Subjects With Grade 3/4 Coagulation Abnormalities
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Subjects With Grade 3/4 Urinalysis Abnormalities
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Subjects With Grade 3/4 Thyroid Function Abnormalities
Description: as for outcome 1
Time Frame: Up to 25 weeks
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue)
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 4, 10, 14, 17, 23, and End of Treatment
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change From Baseline in FACT Kidney Symptom Index Disease-Related Symptoms (FKSI-DRS)
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 4, 10, 14, 17, 23, and End of Treatment
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Diarrhea (FACT-D)
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 4, 10, 14, 17, 23, and End of Treatment
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change From Baseline in Euro Quality of Life - 5 Dimensions (EQ-5D)
Description: as for outcome 1
Time Frame: Baseline, Weeks 1, 4, 10, 14, 17, 23, and End of Treatment
Population: as for outcome 1
Arm/Group | Tivozanib | Sunitinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Collected from the time of signing the Informed Consent Form until 30 days after permanent treatment discontinuation at Week 25 (2 sequential 12-week treatment periods with a 1-week washout period). The Sponsor terminated Study AV-951-12-205 before enrollment was completed, following the negative decision of the US FDA.
Description: Serious treatment-emergent adverse events and treatment-emergent adverse events in Safety (SAF) Population was reported.
Arm/Group | Tivozanib | Sunitinib
Serious Adverse Events (participants affected / at risk) | 6/38 | 7/41
Other Adverse Events (participants affected / at risk) | 35/38 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib (N=38) | Sunitinib (N=41)
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Asthenia (General disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivozanib (N=38) | Sunitinib (N=41)
Diarrhoea (Gastrointestinal disorders) | 17 | 15
Stomatitis (Gastrointestinal disorders) | 8 | 9
Constipation (Gastrointestinal disorders) | 5 | 3
Gingival pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 14
Vomiting (Gastrointestinal disorders) | 3 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Dry mouth (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 10
Flatulence (Gastrointestinal disorders) | 1 | 5
Oral pain (Gastrointestinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 14 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Proteinuria (Renal and urinary disorders) | 1 | 3
Haematuria (Renal and urinary disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 11
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Weight decreased (Investigations) | 4 | 0
Blood creatinine increased (Investigations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Fatigue (General disorders) | 14 | 18
Asthenia (General disorders) | 7 | 9
Oedema peripheral (General disorders) | 3 | 5
Pyrexia (General disorders) | 2 | 5
Hypertension (Vascular disorders) | 19 | 12
Hypotension (Vascular disorders) | 3 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 5 | 1
Dysgeusia (Nervous system disorders) | 4 | 17
Dizziness (Nervous system disorders) | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 2
Chills (General disorders) | 0 | 3
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Neuropathy peripheral (Nervous system disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Lipase increased (Investigations) | 0 | 5
Amylase increased (Investigations) | 0 | 3
Platelet count decreased (Investigations) | 0 | 3
White blood cell count decreased (Investigations) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Eyelid oedema (Eye disorders) | 0 | 3
Jaundice (Hepatobiliary disorders) | 0 | 4
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
The Sponsor terminated Study AV-951-12-205 before enrollment was completed, following the negative decision of the US FDA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No